CLINICAL TRIAL: NCT04553861
Title: Correlation Between Smartwatch-based Blood Pressure Monitoring and Conventional Ambulatory Blood Pressure Monitoring
Brief Title: Smartwatch ABPM vs. Conventional ABPM
Acronym: SamsungWatch
Status: Completed | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Principal Investigator, Young Jin Youn, Assistant Professor, Division of Cardiology, Department of Internal Medicine, Wonju Severance Christian Hospital
Other Study IDs: SamsungWatch
Record Dates: First submitted 2020-09-11; First posted 2020-09-18 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Blood Pressure
Keywords: Blood Pressure; Ambulatory blood pressure monitoring; Smartwatch
MeSH Terms: interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy subjects: Healthy subjects without blood pressure difference on both arm
  Interventions: Device: Ambulatory blood pressure monitoring; Device: Galaxy Watch Active2

INTERVENTIONS:
Device: Ambulatory blood pressure monitoring — Every 30 minutes from 7 AM to 10 PM and every 1 hour from 10 PM to 7 AM
Device: Galaxy Watch Active2 — Every 1 hour by subject (on-demand) from 7 AM to 10 PM and every 5 minutes (automatic) from 10 PM to 7 AM

SUMMARY:
This study aims to investigate the accuracy and precision of the Samsung Smartwatch with conventional ambulatory blood pressure monitoring in healthy volunteers.

DETAILED DESCRIPTION:
Blood pressure (BP) monitoring outside of the medical care environment is an increasingly important part of clinical hypertension assessment and management. Ambulatory BP monitoring (ABPM) uses automatic detection and recording devices for repeated determinations during an extended period, typically 24 hours. This technique has been shown to substantially enhance the clinician's understanding of BP behavior in patients and aid in diagnosis and therapeutic decision making. The ABPM is superior to office BP in predicting target organ, hypertensive cerebrovascular disease, retinopathy, renal abnormalities, and alterations in vascular compliance.1-4) Most of these studies have also demonstrated that a loss of nocturnal decline in BP (so-called non-dipper) conveys excessive risk for stroke and myocardial infarction.

Although conventional ABMP is usually well tolerated by patients, a few problems do exist. A minority of patients do not sleep well with the recorders and tend to have somewhat higher BP values. Cuffs can also rotate, and different arm positions can change BP significantly. Rarely, patients may develop erythema, ecchymoses, petechiae, or superficial phlebitis in the area distal to cuff placement.

Recently, smartwatches that measure BP without a cuff have become available. Since these measurements are relatively more user-friendly than conventional cuff-based measurements, they may aid in more frequent BP monitoring. Currently, only one study compared a non-commercial armband wearable pulse transit time (PTT) system for 24-hour cuff-less BP measurement with ABPM.5) We will investigate the accuracy and precision of Samsung Smartwatch with ABPM in young, healthy volunteers.

ELIGIBILITY:
Inclusion criteria

* Ambulatory healthy subjects
* Subjects aged 20 years or more
* Subjects willing to participate in this study voluntarily Exclusion criteria
* Subjects inability to provide informed consent
* Subjects with any medical history
* Subjects with irregular heart rhythm (e.g. atrial fibrillation, atrial flutter, or bigeminy)
* Subjects unable to wear a watch due to wrist circumference
* Subjects with BP difference 10mmHg or more between left and right arm

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects willing to participate in this trial
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Mean nighttime blood pressure | Baseline
  Correlation of mean nighttime BP between the ABPM and the BP using the smartwatch

SECONDARY OUTCOMES:
Every time point blood pressure | Baseline
  BP differences between the ABPM and the BP using the smartwatch at every time point of measurement
Mean 24-hour blood pressure | Baseline
  Correlation of mean 24-h BP between the ABPM and the BP using the smartwatch
Mean daytime blood pressure | Baseline
  Correlation of mean daytime BP between the ABPM and the BP using the smartwatch
Nighttime dipping | Baseline
  Correlation of nighttime dipping between the ABPM and the BP using the smartwatch
Morning blood pressure | Baseline
  Correlation of morning BP between the ABPM and the BP using the smartwatch

CONTACTS AND LOCATIONS:
Overall Officials: Young Jin Youn, MD, PhD, Principal Investigator — Wonju Severance Christian Hospital
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No